CLINICAL TRIAL: NCT07216040
Title: Harnessing Optimism and Perseverance in the Face of Long COVID~Español (HOPE-LC~Español)
Brief Title: Harnessing Optimism and Perseverance in the Face of Long COVID-Español
Acronym: HOPE-LC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Eric Watson, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-25-01010
Record Dates: First submitted 2025-10-09; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: Post-Acute COVID-19 Syndrome; group therapy; acceptance and commitment therapy; Spanish-speaking
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Single arm pre-post design. Focus is on feasibility with preliminary efficacy as secondary focus.
Masking Description: Single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients Living with Chronic Long-COVID (Experimental): Spanish-speaking patients in the HOPE-LC program.
  Interventions: Behavioral: HOPE-LC~Espanol

INTERVENTIONS:
Behavioral: HOPE-LC~Espanol — 12-week online group therapy program grounded in principles of Acceptance and Commitment Therapy and tailored specifically to living with Long COVID as a chronic condition. HOPE-LC provides community and hope; fostering resilience, adjustment, and critical coping strategies in the face of this debilitating chronic condition.

SUMMARY:
The Harnessing Optimism and Perseverance in the Face of Long COVID (HOPE-LC) program, created by Drs. Eric Watson and Amelia Hicks, is a group therapy model designed to foster resilience, adjustment, and coping skills for those living with chronic Long COVID. HOPE-LC~Español provides a culturally and linguistically adapted version for Spanish-speaking individuals in Queens, developed with input from Spanish-speaking clinicians, Long COVID experts, and people with lived experience. Partnering with H+H/Elmhurst and H+H/Queens, the project aims to recruit 25 participants and evaluate program feasibility and preliminary efficacy.

DETAILED DESCRIPTION:
The Harnessing Optimism and Perseverance in the Face of Long COVID (HOPE-LC) program, developed by Drs. Eric Watson (PI) and Amelia Hicks (co-I), is a 12-week online group therapy program tailored specifically to living with Long COVID as a chronic condition. HOPE-LC provides community and hope; fostering resilience, adjustment, and critical coping strategies in the face of this debilitating chronic condition. Since its inception in 2024, the HOPE-LC groups have engaged 20 patients, emphasizing the need for chronic Long COVID therapeutic interventions.

Through HOPE-LC-Espanol the researchers will translate and adapt the HOPE-LC program into Spanish and expand HOPE-LC's reach to underserved Spanish-speaking communities in Queens and NYC. The aims are: (1) To translate and culturally adapt the HOPE-LC program for Spanish-speaking patients in collaboration with the Advisory Board of Spanish-speaking clinicians, Long COVID experts, and individuals with Long COVID lived experience; (2) In collaboration with the partners at H+H/Elmhurst and H+H/Queens, to conduct targeted recruitment to ensure the researchers are engaging specifically with local Hispanic/Latinx communities in Queens; and (3) To complete the HOPE-LC~Español program for 25 Spanish-speaking individuals experiencing Long COVID within the local Queens community. The researchers will evaluate program feasibility and treatment success to inform future scalability and sustainability as a clinical program.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Speaks and understands Spanish at a level that allows active participation in group-based study procedures.
* Self-reported history of Long COVID/post-COVID condition of any severity or duration, including ongoing emotional or cognitive symptoms affecting daily functioning or a medical professional has diagnosed you with a Long COVID/post-COVID condition of any severity or duration, including ongoing emotional or cognitive symptoms.
* Ability to participate in group sessions either in-person or via telehealth (Zoom).
* Willingness and capacity to provide informed consent.

Exclusion Criteria:

* Presence of severe psychiatric conditions that would preclude participation in group therapy (e.g., active psychosis, suicidal intent requiring immediate intervention).
* Inability to communicate in Spanish sufficiently to engage meaningfully in group sessions.
* Cognitive or physical impairments prevent participation in group sessions or completion of surveys, without available accommodations.
* Concurrent participation in another conflicting interventional trial targeting Long COVID symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Throughout the study period, 12 weeks
  Number of eligible participants screened and enrolled by referral source
Retention rate | Throughout the study period, 12 weeks
  Number of participants completing the intervention (defined as attending at least 8 of 12 sessions)
Number of sessions participants attended | Throughout the study period, 12 weeks
  Feasibility measured via participant attendance
Number of completed surveys | Throughout the study period, 12 weeks
  Feasibility measured via number of surveys completed from participant follow-up and study procedures.
Patient Satisfaction | Post-treatment (Week 12)
  Post-treatment survey assessing participant satisfaction with HOPE-LC~Español. Items are on a 5-point Likert Scale evaluated agreement to statements about their experience in the program (e.g., feeling heard, learning practical strategies, and willingness to recommend the program). The total score range is 5 - 40, with higher ratings indicating greater satisfaction.

SECONDARY OUTCOMES:
DePaul Symptom Questionnaire | Baseline; 6 weeks, 12 weeks
  The DePaul Symptom Questionnaire (DSQ) is a validated tool to assess symptoms, frequency and severity of various symptoms of fatigue and other neurological impairment. Total score range 0-100, with higher scores indicating greater symptom severity and functional impairment.
Brief Illness Perception Questionnaire (BIPQ) | Baseline; 6 weeks, 12 weeks
  The BIPQ assesses cognitive and emotional representations of illness in 8 items + 1 open-ended causal item. Total score range is 0-80, higher scores mean a more negative perception of illness.
Valued Based Living Questionnaire (VLQ) | Baseline; 6 weeks, 12 weeks
  Assesses alignment between personal values and daily actions. Two ratings per domain: (1) Importance (1-10) and (2) Consistency with actions (1-10). Total score range is between 4-40. Higher consistency scores reflect greater valued living (better outcome); lower scores reflect minimal valued living (worse outcome).
Modified COVID-19 Yorkshire Rehabilitation Scale (C19-YRSm) | Baseline; 6 weeks, 12 weeks
  The C19-YRSm is a 17-item self-report scale designed to assess the impact of post-COVID symptoms. Items are rated on a scale from 0 (none of this symptom) to 3 (extremely severe level or impact). The scale includes four subscales:
  Symptom Severity (Questions 1-10; score range: 0-30) Functional Disability (Questions 11-15; score range: 0-15) Other Symptoms (Question 16; score range: 0-25) Overall Health (Question 17; score range: 0-10)
  Full scale from 0-80. Higher scores indicate greater symptom severity and functional impairment.
Patient Health Questionnaire-8 Item (PHQ-8) | Baseline; 6 weeks, 12 weeks
  Patient health questionnaire-8 (PHQ-8) is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. PHQ-8 is an 8-item instrument. Each question is rated on a scale of 0 to 3, total score scale from 0 - 24. Lower scores indicate minimal depression (better outcome) and higher scores indicate severe depression (worse outcome).
Generalized Anxiety Disorder-7 Item (GAD-7) | Baseline; 6 weeks, 12 weeks
  This is a 7-item measure that asks participants to rate the frequency with which they have been bothered by anxiety symptoms within the past two weeks on a scale ranging from 0 ("not at all") to 3 ("nearly every day"). Total scores range from 0-21, with higher scores indicating greater severity of generalized anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Watson, Principal Investigator — Icahn School of Medicine; Amelia Hicks, PhD, Principal Investigator — Icahn School of Medicine
Locations (1):
- Brain Injury Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Proposals should be directed to eric.watson@mountsinai.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third-party website (link to be determined).